CLINICAL TRIAL: NCT02247258
Title: Azathioprine in the Prevention of Ileal Crohn's Disease Postoperative Recurrence: Systematic Versus Endoscopic-directed Treatment. A Multi-center, Randomized, Clinical Practice Evaluation Study.
Brief Title: Azathioprine in the Prevention of Ileal Crohn's Disease Postoperative Recurrence.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: International organization for the study of inflammatory bowel disease (IOIBD) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ML3121
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2014-09

CONDITIONS: Crohn Disease; Recurrence; Azathioprine; Prevention
MeSH Terms: conditions — Crohn Disease; Recurrence | interventions — Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systematic azathioprine group (Active Comparator): Patients randomized to the systematic azathioprine group received 2.0-2.5 mg/kg azathioprine within 14 days from surgery and throughout 102 weeks.
  Interventions: Drug: Azathioprine; Procedure: Ileocolonoscopy; Procedure: Small bowel follow trough
- Endoscopy-driven azathioprine group (Active Comparator): Patients randomized to the endoscopy-driven azathioprine group received no Crohn's disease specific treatment for 26 weeks postoperatively. A first ileocolonoscopy was performed at week 26. In case of endoscopic recurrence (Rutgeerts' score i2 or higher), azathioprine was introduced at a dose of 2.0-2.5 mg/kg until week 102. If not, an ileocolonoscopy was repeated at week 52, and azathioprine started in case of endoscopic recurrence. If no endoscopic recurrence was observed, no Crohn's disease-specific treatment was given until week 102.
  Interventions: Drug: Azathioprine in case of endoscopic recurrence; Procedure: Ileocolonoscopy; Procedure: Small bowel follow trough

INTERVENTIONS:
Drug: Azathioprine — See arm/group descriptions
  Arms: Systematic azathioprine group
Drug: Azathioprine in case of endoscopic recurrence — See arm/group descriptions
  Arms: Endoscopy-driven azathioprine group
Procedure: Ileocolonoscopy — See arm/group descriptions
Procedure: Small bowel follow trough — See arm/group descriptions

SUMMARY:
The objective of this study is to evaluate if in the prevention of postoperative recurrence of ileal Crohn's disease immediate initiation of azathioprine postoperatively is superior to delayed (6- 12 mths.) introduction of azathioprine upon disease recurrence assessed by endoscopic criteria. The primary endpoint, disease recurrence, encompasses symptomatic and surgical recurrence as well as severe endoscopic lesions at the final, 2 year, assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled surgery for Crohn's disease (CD) with ileocolonic resection. Diagnosis of CD confirmed at least 4 months prior to surgery based on radiology and/or endoscopy.
2. Having an increased risk for postoperative relapse for any of the following reasons: (1) active inflammatory disease with C-reactive protein level (CRP) elevated above 10 mg/L, or the use of antibiotics, steroids or biological therapy including infliximab for active ileal disease within 2 months before surgery which were administered for Crohn's disease and not for another unrelated intercurrent inflammatory or infectious disease; (2) perforating disease defined as the presence of entero-enteric or enterocutaneous fistulas or perivisceral abscess formation within 2 months before surgery. Perianal fistulizing disease will not be considered as an indication of perforating disease in the ileum or right-sided colon. (3) Previous ileo-colonic resection, (4) active smoking, (5) age below 30.
3. Males and females 16-75 years old.
4. Curative surgical resection. All macroscopically inflamed colonic segments (except for anorectal involvement) are to be removed at surgery. Stricturoplasties in small bowel segments not involving the anastomotic region are allowed.
5. Patients able to start oral nutrition and oral therapy within 14 days from surgery.
6. Patients able and willing to give written informed consent
7. Women of childbearing potential should have a negative pregnancy test at inclusion.

Exclusion Criteria:

1. Patients who only had strictureplasties or ileal/colonic resection without a new ileo-colonic anastomosis. Patients with ileorectal anastomosis.
2. Patients with no increased risk of postoperative relapse as defined before.
3. Patients with a known intolerance to azathioprine/6-mercaptopurine or with known homozygous thiopurine methyltransferase-low mutation.
4. Patients in whom more than 100 cm of small bowel has been previously resected.
5. Patients with active perianal disease or colorectal stenosis precluding ileocolonoscopy
6. Patients with sepsis or other postoperative complications necessitating use of antibiotics for more than 14 days after surgery.
7. Patients with liver test abnormalities (serum glutamate oxaloacetate transaminase, serum glutamate pyruvate transaminase, alkaline phosphatase, bilirubin > 2 ULN), leucopenia (<3000 white blood cell count /µL, <1500 neutrophils /µL), thrombopenia with < 50.000 platelets/mm3.
8. Patients with severe renal, pulmonary or cardiac disease.
9. Pregnant or lactating women.
10. Ongoing alcohol or substance abuse.
11. Ongoing or recent (within 6 months) infectious disease (viral hepatitis, tuberculosis, AIDS, Herpes zoster related disease).
12. Known malignancy 5 years from surgery except for superficial epithelioma of the skin with curative resection.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-10; Primary Completion 2014-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Endoscopic remission | Week 102
  The proportion of patients with endoscopic remission (Rutgeerts' postoperative endoscopic score i0 or i1) at 102 weeks

SECONDARY OUTCOMES:
Complete endoscopic remission | Week 102
  The percentage of patients with a Rutgeerts' score of i0 at 102 weeks
Absence of endoscopic relapse | Week 102
  The percentage of patients with a Rutgeerts' score of i0-i2 at 102 weeks
Clinical remission | Week 102
  The percentage of patients in clinical remission (Crohn's disease activity index, CDAI <150) at 102 weeks
Sustained clinical remission | Week 102
  Crohn's disease activity index, CDAI < 150 throughout the 102 weeks study period
Radiological remission | Week 102
  The percentage of patients with radiological remission at 102 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gert Van Assche, MD PhD, Principal Investigator — UZ Leuven
Locations (4):
- Belgium (2):
  - Imelda Ziekenhuis, Bonheiden
  - UZ Leuven, Leuven
- Univerzity Karlovy, Prague, Czechia
- Evangelismos Hospital, Athens, Greece

REFERENCES:
- [Derived] Ferrante M, Papamichael K, Duricova D, D'Haens G, Vermeire S, Archavlis E, Rutgeerts P, Bortlik M, Mantzaris G, Van Assche G; International Organization for Study of Inflammatory Bowel Diseases. Systematic versus Endoscopy-driven Treatment with Azathioprine to Prevent Postoperative Ileal Crohn's Disease Recurrence. J Crohns Colitis. 2015 Aug;9(8):617-24. doi: 10.1093/ecco-jcc/jjv076. Epub 2015 Apr 29. PMID 25926532